CLINICAL TRIAL: NCT01864226
Title: A Single-Center, Randomized, Investigator/Subject-Blind, Adaptive Multiple Ascending-Dose, Placebo-Controlled, Parallel Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of RO5545965 Following Oral Administration in Healthy Subjects.
Brief Title: A Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of RO5545965 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: BP28845
Record Dates: First submitted 2013-05-24; First posted 2013-05-29 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo
- RO5545965 (Experimental)
  Interventions: Drug: RO5545965

INTERVENTIONS:
Drug: RO5545965 — Multiple ascending doses
  Arms: RO5545965
Drug: placebo — Multiple ascending doses
  Arms: Placebo

SUMMARY:
This single-center, randomized, investigator/subject-blind, adaptive multiple ascending-dose, placebo-controlled study will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of RO5545965 in healthy volunteers. Subjects will be randomized to receive either RO5545965 or matching placebo daily for 12 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female volunteers, 18 - 64 years of age, inclusive Healthy status is defined by absence of evidence of any active or chronic disease following detailed medical and surgical history and a complete physical examination
* Body mass index (BMI) 18 to 30 kg/m2 inclusive
* Female subject must be post-menopausal or surgically sterile
* Male subjects with female partners of child-bearing potential must use two methods of contraception, one of which must be a barrier method, for the duration of the study and for at least 30 days after the last dose of study drug

Exclusion Criteria:

* History of any clinically significant disease or disorder
* Concomitant disease or condition that could interfere with, or the treatment of which might interfere with, the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
* Clinically significant abnormalities in laboratory test results
* Suspicion of regular consumption of drug of abuse
* Positive for hepatitis B, hepatitis C or HIV infection
* Participation in an investigational drug or device study within 90 days prior to screening
* Regular smoker (>5 cigarettes, >1 pipeful or >1 cigar per day)
* History of clinically significant hypersensitivity or allergic drug reactions

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2013-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | approximately 3 months

SECONDARY OUTCOMES:
Pharmacokinetics: Area under the concentration-time curve (AUC) | 17 days
Pharmacokinetics: Plasma concentrations | 17 days
Pharmacokinetics: Urine concentrations | 13 days
Pharmacodynamics: Serum prolactin levels | Day 12
Pharmacodynamics: Glucose tolerance test | Day 11
Pharmacodynamics: Probabilistic learning tasks | Days 6, 8 and 10

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Zuidlaren, Netherlands